CLINICAL TRIAL: NCT07104890
Title: Evaluation of Enhanced Recovery After Surgery (ERAS) Protocol on Postoperative Recovery in Elective Cesarean Sections
Brief Title: Enhanced Recovery After Surgery (ERAS) Protocol in Elective Cesarean Sections
Acronym: ERAS-CS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Havva Betül Bacak (Other Government)
Responsible Party: Sponsor-Investigator, Havva Betül Bacak, M.D, Gaziosmanpasa Research and Education Hospital
Organization: Gaziosmanpasa Research and Education Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOEAH-ERAS-CS01
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Elective Cesarean Section; Postoperative Recovery; Enhanced Recovery After Surgery (ERAS)
Keywords: Cesarean Section; Elective Cesarean; Enhanced Recovery After Surgery; ERAS; Postoperative Recovery; Early Mobilization; Postoperative Pain; Multimodal Analgesia; Obstetric Surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Enhanced Recovery After Surgery; Clinical Protocols; Early Ambulation

STUDY DESIGN:
Intervention Model Description: This is a single-center, prospective, randomized, parallel-group clinical trial.
  Participants were randomly assigned in a 1:1 ratio to either the ERAS protocol group or the standard care control group.
  Both groups were followed concurrently for postoperative recovery outcomes after elective cesarean section.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS Protocol Group (Experimental): Participants in this arm will receive the Enhanced Recovery After Surgery (ERAS) protocol during elective cesarean section. The ERAS protocol includes early oral intake, early mobilization, opioid-sparing multimodal analgesia, prophylactic antiemetics, early urinary catheter removal, and gum chewing to stimulate bowel function. Postoperative outcomes such as breastfeeding initiation, gas passage, oral intake time, mobilization, and VAS pain scores will be evaluated.
  Interventions: Behavioral: Enhanced Recovery After Surgery (ERAS) Protocol, which includes early oral intake, early mobilization, opioid-sparing multimodal analgesia, prophylactic antiemetics, early urinary catheter removal, an
- Standard Care Group (Active Comparator): Participants in this arm will receive standard perioperative cesarean care, which includes overnight fasting, delayed oral intake until gas passage, routine analgesia with paracetamol, NSAIDs and opioids as needed, later urinary catheter removal, and routine postoperative mobilization. Outcomes will be assessed similarly to the ERAS group.
  Interventions: Behavioral: Enhanced Recovery After Surgery (ERAS) Protocol, which includes early oral intake, early mobilization, opioid-sparing multimodal analgesia, prophylactic antiemetics, early urinary catheter removal, an

INTERVENTIONS:
Behavioral: Enhanced Recovery After Surgery (ERAS) Protocol, which includes early oral intake, early mobilization, opioid-sparing multimodal analgesia, prophylactic antiemetics, early urinary catheter removal, an — The Enhanced Recovery After Surgery (ERAS) Protocol for elective cesarean section includes a multimodal perioperative care approach aimed at accelerating postoperative recovery. Key components are early oral intake, early mobilization, opioid-sparing multimodal analgesia, prophylactic antiemetics, early removal of the urinary catheter, and gum chewing to stimulate bowel function. This protocol is compared with Standard Perioperative Cesarean Care, which involves overnight fasting, delayed oral intake until bowel function returns, conventional analgesia, later mobilization, and routine catheter removal.

SUMMARY:
This study evaluates the effect of the Enhanced Recovery After Surgery (ERAS) protocol on early postoperative recovery in women undergoing elective cesarean section.

Eighty-four pregnant women, aged 18 years or older, at 37 weeks of gestation or beyond, without chronic medical conditions, and classified as ASA I-II, were enrolled. Participants were randomly assigned to either:

ERAS group - received the ERAS protocol, including early oral intake, early mobilization, multimodal analgesia, and enhanced perioperative care

Control group - received standard perioperative cesarean section care

The study compared breastfeeding initiation time, gas passage, oral intake, mobilization time, and postoperative pain scores (VAS) between the two groups.

The aim is to determine whether ERAS can accelerate recovery, reduce pain, and improve maternal comfort after elective cesarean delivery.

DETAILED DESCRIPTION:
Enhanced Recovery After Surgery (ERAS) protocols aim to accelerate postoperative recovery, reduce complications, and shorten hospital stays. While ERAS has been widely implemented in general and gynecologic surgeries, its application in obstetric surgery, particularly elective cesarean delivery, remains limited.

This single-center, prospective, randomized clinical trial was conducted at the University of Health Sciences, Istanbul Gaziosmanpasa Training and Research Hospital, between October 2022 and December 2022. Eighty-four women scheduled for elective cesarean section were enrolled. Eligible participants were 18 years or older, at ≥37 weeks of gestation, ASA I-II, without chronic comorbidities, and provided written informed consent.

Participants were randomized (1:1) into two groups:

ERAS group: Managed with ERAS protocol including early oral intake, early mobilization, multimodal analgesia with opioid-sparing strategies, prophylactic antiemetics, early urinary catheter removal, and gum chewing to stimulate bowel function.

Control group: Managed with standard perioperative cesarean care including delayed oral intake, standard pain management, and later mobilization.

Primary outcomes included breastfeeding initiation time, gas passage, time to oral intake, mobilization time, and postoperative pain scores (VAS at 24 and 48 hours). Secondary outcomes included nausea-vomiting incidence and overall postoperative recovery profile.

The study aims to determine whether ERAS protocols improve postoperative recovery and patient comfort after elective cesarean section and to support the implementation of ERAS as a standard in obstetric surgery.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women aged 18 years or older

Gestational age ≥37 weeks

Classified as ASA I or ASA II

Scheduled for elective cesarean section under spinal anesthesia

Able and willing to provide informed consent

No chronic systemic diseases

Exclusion Criteria:

Age <18 years

Gestational age <37 weeks

Emergency cesarean delivery

ASA III or higher

Presence of obstetric complications (e.g., preeclampsia, placenta previa, placental abruption, fetal distress)

Chronic comorbidities (e.g., diabetes, hypertension, cardiac or pulmonary disease)

Declines spinal anesthesia or unable to provide consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only biologically female participants who are pregnant and scheduled for elective cesarean section are eligible for the study. Self-identified gender does not alter eligibility; participants must be biologically female.
Enrollment: 84 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Time to First Mobilization After Cesarean Section | Within 24 hours postoperatively
  Time from the end of elective cesarean section surgery to the patient's first ambulation, measured in hours. Early mobilization reflects enhanced postoperative recovery and is a key indicator of the ERAS protocol's effectiveness.

SECONDARY OUTCOMES:
Incidence of Postoperative Nausea and Vomiting | Within 48 hours postoperatively
  Assessment of the presence and duration of postoperative nausea and vomiting (PONV) following elective cesarean section. Nausea and vomiting episodes will be recorded and analyzed to compare the incidence between the ERAS protocol group and the standard care group.

CONTACTS AND LOCATIONS:
Locations (1):
- Bartın City Hospital, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study is single-center, involves a small sample size of 84 participants, and contains sensitive obstetric patient information. Only de-identified summary data will be reported in publications.

REFERENCES:
- [Background] Khalafallah AM, Susic N, Shah KH, Knott MV, Berke CN, Gurses ME, Lu VM, Ivan ME, Komotar RJ, Shah AH. Evaluating safety and feasibility of same-day discharge after laser interstitial thermal therapy: a pilot study with a matched control group. J Neurooncol. 2025 Sep;174(2):341-347. doi: 10.1007/s11060-025-05055-4. Epub 2025 May 12. PMID 40355785
- [Background] Zhang X, Ruan Y, Yuan Y, Li K. Is it necessary to maintain high adherence to enhanced recovery after surgery (ERAS) protocols?-A systematic review and meta-analysis. Curr Probl Surg. 2025 Aug;69:101814. doi: 10.1016/j.cpsurg.2025.101814. Epub 2025 May 30. No abstract available. PMID 40716849